CLINICAL TRIAL: NCT04425538
Title: A Phase 2 Trial of Infliximab in Coronavirus Disease 2019 (COVID-19).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000564
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Results first posted 2021-12-03 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Infliximab (Experimental): All patients enrolled into this trial will be assigned to the Infliximab arm. Patients will be treated with infliximab on Day 1, and may be re-treated per protocol and at the discretion of the investigator.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Either infliximab or infliximab-abda will be used at the discretion of the investigator
  Other Names: infliximab-abda

SUMMARY:
The investigators hypothesize that early institution of TNFα inhibitor therapy in patients with severe COVID-19 infections will prevent further clinical deterioration and reduce the need for advanced cardiorespiratory support and early mortality. To address this hypothesis, a prospective, single center, phase 2 trial is proposed to assess the efficacy of infliximab or infliximab-abda in hospitalized adult patients with severe or critical COVID-19. Observations from this study will inform the conduct of prospective randomized controlled studies to follow.

DETAILED DESCRIPTION:
The investigators hypothesize that early institution of TNFα inhibitor therapy in patients with severe COVID-19 infections will prevent further clinical deterioration and reduce the need for advanced cardiorespiratory support and early mortality. To address this hypothesis, a prospective, single center, phase 2 trial is proposed to assess the efficacy of infliximab or infliximab-abda in hospitalized adult patients with severe or critical COVID-19. Observations from this study will inform the conduct of prospective randomized controlled studies to follow.

Infliximab and Infliximab-abda are TNFα inhibitors currently FDA-approved for the treatment of autoimmune disorders, including Crohn's disease and rheumatoid arthritis. The risks and adverse reactions are described in the approved prescribing information for infliximab (or infliximab-abda). Infliximab will be used when available. Should infliximab be unavailable in the pharmacy, infliximab-abda, a biosimilar, will be used.

Treatment with infliximab or infliximab-abda 5mg/kg IV should ideally be administered within 6 hours of enrollment, and no more than 24 hours following enrollment. Pre-medication with Tylenol 650 mg once 30 minutes prior to infusion would be recommended. Other pre-medications may be given at the discretion of the treating physician. These include diphenhydramine 50mg by mouth, as well as prednisone 20mg by mouth, both given 30 minutes prior to infusion. Pulse and blood pressure should be monitored every 30 minutes during the infusion, and patients should be monitored for at least 30 minutes following the infusion.

Retreatment with infliximab is permitted at treating physician discretion 7-21 days following primary therapy and based on initial response; the usual treatment schedule is every 2 weeks, this interval is not strictly enforced given the uncertainty of outcomes with primary therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Able to provide informed consent
3. Hospitalized adult patients with pneumonia evidenced by chest X-ray or CT scan
4. Laboratory (RT-PCR) confirmed infection with 2019-nCoV or strongly suspected to be infected with SARS-COV2 with confirmation studies pending
5. And at least one of the following:

   1. Respiratory frequency ≥30/min
   2. Blood oxygen saturation ≤93% on RA
   3. Partial pressure of arterial oxygen to fraction of inspired oxygen ratio (PaO2/FiO2) <300
   4. Worsening of lung involvement, defined as an increase in number and/or extension of pulmonary areas of consolidation, need for increased FiO2 to maintain stable O2 saturation, or worsening O2 saturation of >3% with stable FiO2

Exclusion Criteria:

1. Treatment with any TNFα inhibitor in the past 30 days
2. Known hypersensitivity to any TNFα inhibitor, murine proteins, or any component of the formulation
3. Presence of any of the following abnormal laboratory values at screening: absolute neutrophil count (ANC) less than 1000 mm3, hemoglobin <8.0g/L, platelets <50,000 per mm3, or AST or ALT greater than 5 x ULN
4. Known active or latent Hepatitis B
5. Known or suspected active tuberculosis (TB) or a history of incompletely treated or latent TB.
6. Pregnancy
7. Intubated for >48hours
8. Patients with uncontrolled systemic bacterial or fungal infections (Patients with a history of positive bacterial or fungal cultures but on enrollment are on appropriate therapy with negative repeat cultures may be enrolled)
9. Serious co-morbidity, including:

   1. Myocardial infarction (within last month)
   2. Moderate or severe heart failure (New York Heart Association (NYHA) class III or IV)
   3. Acute stroke (within last month)
   4. Uncontrolled malignancy
   5. Stage 4 severe chronic kidney disease or requiring dialysis (i.e. estimated glomerular filtration rate (eGFR) < 30 ml /min/1.73 m^2) at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mathew, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hachem H, Godara A, Schroeder C, Fein D, Mann H, Lawlor C, Marshall J, Klein A, Poutsiaka D, Breeze JL, Joshi R, Mathew P. Rapid and sustained decline in CXCL-10 (IP-10) annotates clinical outcomes following TNF-alpha antagonist therapy in hospitalized patients with severe and critical COVID-19 respiratory failure. medRxiv [Preprint]. 2021 Jun 2:2021.05.29.21258010. doi: 10.1101/2021.05.29.21258010. PMID 34100026
- [Result] Hachem H, Godara A, Schroeder C, Fein D, Mann H, Lawlor C, Marshall J, Klein A, Poutsiaka D, Breeze JL, Joshi R, Mathew P. Rapid and sustained decline in CXCL-10 (IP-10) annotates clinical outcomes following TNFalpha-antagonist therapy in hospitalized patients with severe and critical COVID-19 respiratory failure. J Clin Transl Sci. 2021 Jun 25;5(1):e146. doi: 10.1017/cts.2021.805. eCollection 2021. PMID 34457357

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infliximab
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Age, Customized [Count of Participants; unit: Participants]
  18-40 years | 1
  41-60 years | 7
  >60 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 4
  Black/African American | 2
  Chinese | 3
  Other Asian | 2
  Hispanic/Latino | 4
  Other | 1
  Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Time to Improvement in Oxygenation
Description: Time to improvement in oxygenation (increase in SpO2/FiO2 of 50 or greater compared to the baseline SpO2/FiO2)
Time Frame: 28 Days
Population: 15 patients met this endpoint whereby duration data could be obtained
Measure: Median (Full Range); unit: Days
Arm/Group | Infliximab
Number analyzed (Participants) | 15
Days | 4 [1 to 12]

2. Primary Outcome: Number of p[Atients With Improvement in Oxygenation
Description: Number of participants who showed improvement in oxygenation (increase in SpO2/FiO2 of 50 or greater compared to the baseline SpO2/FiO2)
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Participants | 15

3. Secondary Outcome: 28-Day Survival Status
Description: Number of patients who were confirmed to be alive 28 days from enrollment onto the study.
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Participants | 15

4. Secondary Outcome: Duration of Supplemental Oxygen Administration by Nasal Cannula
Description: Duration of supplemental oxygen administration by nasal cannula, simple face mask, or other similar oxygen delivery device
Time Frame: 28 Days
Measure: Median (Full Range); unit: Days
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Days | 3 [1 to 4]

5. Secondary Outcome: Duration of Non-invasive Ventilation or by Non-rebreather Mask or High-flow Nasal Cannula
Description: Duration of non-invasive ventilation or by non-rebreather mask or high-flow nasal cannula
Time Frame: 28 Days
Measure: Median (Full Range); unit: Days
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Days | 2.5 [2 to 6]

6. Secondary Outcome: Number of Patients Requiring Mechanical Ventilation
Description: Number of patients enrolled who required mechanical ventilation
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Participants | 7

7. Secondary Outcome: Number of Patients Requiring Vasopressor Support
Description: Number of participants who required vasopressor support
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Participants | 3

8. Secondary Outcome: Number of Patients Requiring Extracorporeal Membrane Oxygenation
Description: Number of patients requiring extracorporeal membrane oxygenation
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Participants | 1

9. Secondary Outcome: Number of Patients With Fever
Description: Number of patients who exhibited fever during the study period
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Participants | 12

10. Secondary Outcome: Correlation of Dynamic Changes in IP-10 to Cytokine Profile
Description: Correlation of dynamic changes in IP-10 to cytokine profile between day 3 and baseline
Time Frame: 3 Days
Measure: Number; unit: Correlation coefficient
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Correlation coefficient
  CXCL9 | 0.652
  IL-15 | 0.605
  FLT-3L | 0.601
  IL-12p40 | 0.585
  IL-3 | .571
  M-CSF | 0.564
  MDC | 0.528
  IFN-A2 | 0.509
  IL-5 | .501
  IL-18 | .484

11. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization
Time Frame: 28 Days
Measure: Median (Full Range); unit: days
Arm/Group | Infliximab
Number analyzed (Participants) | 17
days | 8 [1 to 28]

12. Secondary Outcome: Number of Patients Who Developed Secondary Infections
Description: Number of patients who developed secondary infections
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Participants | 7

13. Secondary Outcome: Number of Patients Requiring Supplemental Oxygen Administration by Nasal Cannula
Description: Incidence of supplemental oxygen administration by nasal cannula, simple face mask, or other similar oxygen delivery device
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Participants | 14

14. Secondary Outcome: Duration of Mechanical Ventilation
Description: duration of use of mechanical ventilation (for patients requiring mechanical ventilation)
Time Frame: 28 Days
Population: 7 of 17 enrolled patients required mechanical ventilation
Measure: Median (Full Range); unit: days
Arm/Group | Infliximab
Number analyzed (Participants) | 7
days | 10 [5 to 28]

15. Secondary Outcome: Number of Patients Requiring Non-invasive Ventilation or by Non-rebreather Mask or High-flow Nasal Cannula
Description: Number of participants who required non-invasive ventilation or by non-rebreather mask or high-flow nasal cannula
Time Frame: 28 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 17
Participants | 8

16. Secondary Outcome: Assessment of Cytokine and Inflammatory Profile at Baseline
Description: Assessment of cytokine and inflammatory profile at baseline (TNFα, IL-1b, IL-2, IL-6, ferritin) after therapy
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Infliximab
Number analyzed (Participants) | 17
ng/mL
  TNFα | 109.2 (53.4)
  IL-1β | 42.3 (97.8)
  IL-2 | 1.46 (2.21)
  IL-6 | 69.2 (130.85)
  Ferritin | 1972.12 (1517.56)

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected for each patient beginning at the time of first infliximab dose through 28 days following the last dose of infliximab. Study-wide, adverse event collection was conducted for approximately 8 months.
Description: Serious adverse events and all-cause mortality were collected according to clinicaltrials.gov definitions. For other adverse events, only adverse events of special interest were collected for the purposes of this trial. Adverse events of special interest include infusion reactions from infliximab treatment, anaphylaxis, and any other event deemed by the investigator to be directly related to infliximab treatment.
Arm/Group | Infliximab
All-Cause Mortality (participants affected / at risk) | 2/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=17)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Covid-Associated Pulmonary Aspergillosis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab (N=17)
AST Elevation (Investigations) | 9
ALT Elevation (Investigations) | 8
Acute Infusion Reaction (General disorders) | 2
Lung Infection (Infections and infestations) | 8
Hyperglycemia (Investigations) | 1
Acute Kidney Injury (Renal and urinary disorders) | 3
Herpes Simplex Reactivation (Infections and infestations) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Intermittent Sinus Bradycardia (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT04425538/Prot_SAP_000.pdf